CLINICAL TRIAL: NCT04470427
Title: A Phase 3, Randomized, Stratified, Observer-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Immunogenicity of mRNA-1273 SARS-CoV-2 Vaccine in Adults Aged 18 Years and Older
Brief Title: A Study to Evaluate Efficacy, Safety, and Immunogenicity of mRNA-1273 Vaccine in Adults Aged 18 Years and Older to Prevent COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1273-P301; 75A50120C00034 (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2020-07-11; First posted 2020-07-14 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A is observer-blind. Part B is open-label; participants can request to be unblinded by scheduling a Participant Decision clinic visit. Part C offers participants the option to receive a booster dose for those participants who received at least one dose of mRNA-1273 in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1273 (Experimental): Part A (Blinded): Participants will receive 1 intramuscular (IM) injection of 100 microgram (μg) mRNA-1273 on Day 1 and on Day 29.
  Part B (Open-label): Participants who receive mRNA-1273-matching placebo during Part A and choose to be unblinded by participating in Part B, will receive 1 IM injection of 100 μg mRNA-1273 on Day 1 and Day 29. Participants who are only able to receive 1 dose of mRNA-1273 due to administrative reasons, will receive 1 IM injection of 100 μg mRNA-1273 on Day 1, if the participant chooses.
  Part C: Eligible participants in Part B who choose to receive booster dose of mRNA-1273, will receive 1 IM injection of 50 μg mRNA-1273 on Day 1.
  Interventions: Biological: mRNA-1273; Biological: Placebo
- Placebo (Placebo Comparator): Part A only: Participants will receive 1 IM injection of mRNA-1273-matching placebo on Day 1 and on Day 29, if the participant chooses.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: mRNA-1273
Biological: Placebo — 0.9% sodium chloride (normal saline) injection

SUMMARY:
The mRNA-1273 vaccine is being developed to prevent COVID-19, the disease resulting from Severe Acute Respiratory Syndrome coronavirus (SARS-CoV-2) infection. The study is designed to primarily evaluate the efficacy, safety, and immunogenicity of mRNA-1273 to prevent COVID-19 for up to 2 years after the second dose of mRNA-1273.

DETAILED DESCRIPTION:
This is a 3-part Phase 3 study, with Part A (Blinded Phase), Part B (Open-label Observational Phase), and Part C (Booster Dose Phase). Participants in Part A are blinded to their treatment assignment, with participants receiving either mRNA-1273 vaccine or placebo. Part B of the study is designed to offer participants to be unblinded so that participants who received placebo in Part A can request 2 doses of open-label mRNA-1273 vaccine. Additionally, participants who choose to be unblinded and were only able to receive 1 dose of mRNA-1273 due to administrative reasons, can choose to receive the second dose of mRNA-1273 during Part B. In Part C, a booster dose will be provided for all eligible participants who choose to receive one.

Please access www.modernatx.com/cove-study for additional information, such as Study Overview, Participation, and Site Locations along with contact numbers for each location for the study.

ELIGIBILITY:
Inclusion Criteria:

* (Part A only) Participants who are at high risk of SARS-CoV-2 infection, defined as adults whose locations or circumstances put them at appreciable risk of exposure to SARS-CoV-2 and COVID-19.
* Understands and agrees to comply with the study procedures and provides written informed consent.
* Able to comply with study procedures based on the assessment of the Investigator.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal (defined as amenorrhea for ≥12 consecutive months prior to Screening without an alternative medical cause). A follicle-stimulating hormone (FSH) level may be measured at the discretion of the Investigator to confirm postmenopausal status.
* Female participants of childbearing potential may be enrolled in the study if the participant fulfills all the following criteria:

  * Has a negative pregnancy test at Screening and on the day of the first dose (Day 1, open-label Day 1, and booster dose Day 1).
  * Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose (Day 1).
  * Has agreed to continue adequate contraception through 3 months following the last dose (Day 29, open-label Day 29, and booster dose Day 1).
  * Is not currently breastfeeding.
* Healthy adults or adults with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
* (Part C Only) Is currently enrolled in Part B of the current study (mRNA-1273-P301).
* (Part C Only) Has received at least 1 dose of mRNA-1273 in the current study (mRNA-1273-P301).

Exclusion Criteria:

* Is acutely ill or febrile 72 hours prior to or at Screening or dosing (Part B and Part C). Fever is defined as a body temperature ≥38.0°Celsius/100.4°Fahrenheit. Participants meeting this criterion may be rescheduled within the relevant window periods. Afebrile participants with minor illnesses can be enrolled/dosed at the discretion of the Investigator.
* Is pregnant or breastfeeding.
* (Part A Only) Known history of SARS-CoV-2 infection.
* Prior (Part A) or concurrent (Part B and Part C) administration of non-study coronavirus (SARS-CoV, Middle East Respiratory Syndrome [MERS]-CoV) vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19.
* (Part A Only) Demonstrated inability to comply with the study procedures.
* An immediate family member or household member of this study's personnel.
* Known or suspected allergy or history of anaphylaxis, urticaria, or other significant adverse reaction to the vaccine or its excipients.
* Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
* Has received or plans to receive a vaccine within 28 days prior to the first dose (Day 1) or plans to receive a non-study vaccine within 28 days prior to or after any dose of investigational product (IP) (except for seasonal influenza vaccine).
* (Part A only) Has participated in an interventional clinical study within 28 days prior to the day of enrollment.
* Immunosuppressive or immunodeficient state, including human immunodeficiency virus (HIV) infection, asplenia, and recurrent severe infections.
* Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to IP dose administration (for corticosteroids ≥20 milligram (mg)/day of prednisone equivalent).
* Has received systemic immunoglobulins or blood products within 3 months prior to the day of IP dose administration.
* Has donated ≥450 milliliters (mL) of blood products within 28 days prior to IP dose administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30415 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (100):
- United States (100):
  - Ascension St. Vincent Birmingham, Birmingham, Alabama
  - Synexus Clinical Research US, Inc. - Birmingham, Birmingham, Alabama
  - Hope Research Institute, Chandler, Arizona
  - Synexus Clinical Research US, Inc. - Phoenix West, Glendale, Arizona
  - Hope Research Institute, Peoria, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Quality of Life Medical and Research Center, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Advanced Clinical Research - Rancho Paseo, Banning, California
  - University of California San Diego, La Jolla, California
  - eStudySite - La Mesa, La Mesa, California
  - UCLA Vine Street Clinic CRS, Los Angeles, California
  - VA Greater Los Angeles Healthcare (veterans only), Los Angeles, California
  - Paradigm Clinical Research Institute Inc, Redding, California
  - Benchmark Research - Sacramento, Sacramento, California
  - Medical Center For Clinical Research - M3 Wake Research, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Lynn Institute of The Rockies, Colorado Springs, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Accel Research Site, DeLand, Florida
  - Research Centers of America, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Synexus - Optimal Research - Melbourne, Melbourne, Florida
  - Suncoast Research Group, Miami, Florida
  - University of Miami, Miami, Florida
  - Synexus Clinical Research US, Inc. - Orlando, Orlando, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Grady Health System, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Hope Clinic of The Emory Vaccine Center, Decatur, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Synexus Clinical Research US, Inc. - Chicago, Chicago, Illinois
  - UIC Project WISH CRS, Chicago, Illinois
  - University of Chicago-Hospital, Chicago, Illinois
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Alliance for Multispecialty Research, Newton, Kansas
  - Alliance for Multispecialty Research- East Wichita, Wichita, Kansas
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Benchmark Research - Metairie, Metairie, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Synexus - Optimal Research - Rockville, Rockville, Maryland
  - Meridian Clinical Research, Rockville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - MediSync Clinical Research Hattiesburg Clinic, Petal, Mississippi
  - Saint Louis University, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, Grand Island, Nebraska
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New Jersey Medical School, Newark, New Jersey
  - Meridian Clinical Research, Binghamton, New York
  - Weill Cornell Chelsea - (CRS), New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Tryon Medical Partners, Charlotte, North Carolina
  - Carolina Institute for Clinical Research - M3 Wake Research, Fayetteville, North Carolina
  - M3 Wake Research, Inc - M3 Wake, Raleigh, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Synexus Clinical Research US, Inc. - Cincinnati, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Cincinnati CRS, Cincinnati, Ohio
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Crisor, Medford, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC University Center, Pittsburgh, Pennsylvania
  - Keystone VitaLink Research, Anderson, South Carolina
  - Keystone VitaLink Research - Greenville, Greenville, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Keystone VitaLink Research - Spartanburg, Spartanburg, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - WR-ClinSearch, Chattanooga, Tennessee
  - Alliance for Multispecialty Research, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Medical Arts Building, Nashville, Tennessee
  - Vanderbilt University Medical Center, Medical Center North, Nashville, Tennessee
  - Benchmark Research - Austin, Austin, Texas
  - Synexus - Optimal Research - Austin, Austin, Texas
  - Tekton Research, Austin, Texas
  - Advanced Clinical Research - Be Well MD, Cedar Park, Texas
  - Global Medical Research - M3 Wake Research, Dallas, Texas
  - Synexus Clinical Research US, Inc. - Dallas, Dallas, Texas
  - Benchmark Research - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - DM Clinical Research - Texas Center For Drug Development, Houston, Texas
  - Laguna Clinical Research, Laredo, Texas
  - Centex Studies, McAllen, Texas
  - Benchmark Research - San Angelo, San Angelo, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Synexus Clinical Research US, Inc. - Salt Lake City, Murray, Utah
  - Foothill Family Clinic - North, Salt Lake City, Utah
  - Foothill Family Clinic-South Clinic, Salt Lake City, Utah
  - Kaiser Permanente - Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaplonek P, Bertera H, Lee DW, Cizmeci D, Yu WH, Wu K, Chalkias S, Wahid R, Edwards D, Alter G, Henry C. IgG4 Neutralization and Sustained Total IgG Fc-Effector Functions Following Repeated SARS-CoV-2 Vaccination with mRNA-1273. Infect Dis Ther. 2026 Feb 1. doi: 10.1007/s40121-026-01303-w. Online ahead of print. PMID 41622397
- [Derived] Kenny A, van der Laan L, Gilbert P, Carone M. Inference on Controlled Effects for Assessing Immune Correlates of Protection Based on a Cox Model. Stat Med. 2025 Dec;44(28-30):e70347. doi: 10.1002/sim.70347. PMID 41369204
- [Derived] Ashby E, Janes H, Follmann D, Gilbert PB, Zhou H, Wang X, Girard B, Priddy F, Kublin JG, Corey L, Neuzil KM, Baden LR, El Sahly HM, Zhang B; COVE study group. Validating and leveraging non-SARS-CoV-2 respiratory infection as a negative control outcome in a phase 3 COVID-19 vaccine trial with extended observational follow-up. Am J Epidemiol. 2026 Jan 8;195(1):168-177. doi: 10.1093/aje/kwaf176. PMID 40838594
- [Derived] Follmann D, Wang X, Baden LR, El Sahly HM, Essink B, Gilbert P, Janes HE, Kelley CF, Berman MA, Frank I, Chu E, Deng W, Priddy F, Dixit A, Tomassini JE, Das R, Miller J, Zhou H. Who to Boost When: The Effect of Age and Dosing Interval on Delta and Omicron COVID-19 Incidence in the Open-label Phase of the COVE Trial. Open Forum Infect Dis. 2024 Nov 25;11(12):ofae689. doi: 10.1093/ofid/ofae689. eCollection 2024 Dec. PMID 39679349
- [Derived] Zhang B, Fong Y, Fintzi J, Chu E, Janes HE, Kenny A, Carone M, Benkeser D, van der Laan LWP, Deng W, Zhou H, Wang X, Lu Y, Yu C, Borate B, Chen H, Reeder I, Carpp LN, Houchens CR, Martins K, Jayashankar L, Huynh C, Fichtenbaum CJ, Kalams S, Gay CL, Andrasik MP, Kublin JG, Corey L, Neuzil KM, Priddy F, Das R, Girard B, El Sahly HM, Baden LR, Jones T, Donis RO, Koup RA, Gilbert PB, Follmann D; United States Government (USG) COVID-19 Immune Assays Team; Moderna, Inc. Team; Coronavirus Vaccine Prevention Network (CoVPN)/Coronavirus Efficacy (COVE) Team; USG/CoVPN Biostatistics Team. Omicron COVID-19 immune correlates analysis of a third dose of mRNA-1273 in the COVE trial. Nat Commun. 2024 Sep 11;15(1):7954. doi: 10.1038/s41467-024-52348-9. PMID 39261482
- [Derived] Janes H, Fisher LH, Kee JJ, Parameswaran L, Goepfert PA, Falsey AR, Ludwig J, Magaret CA, Gilbert PB, Kublin JG, Rouphael N, Sobieszczyk ME, El Sahly HM, Baden LR, Grinsztejn B, Walsh SR, Gray GE, Kotloff KL, Gay CL, Greninger AL, Tapia MD, Hammershaimb EA, Priddy FH, Green JA, Struyf F, Dunkle L, Neuzil KM, Corey L, Huang Y. Association Between SARS-CoV-2 Viral Load and COVID-19 Vaccination in 4 Phase 3 Trials. J Infect Dis. 2024 Dec 16;230(6):1384-1389. doi: 10.1093/infdis/jiae400. PMID 39225478
- [Derived] Turley CB, Tables L, Fuller T, Sanders LJ, Scott H, Moodley A, Woodward Davis A, Leav B, Miller J, Schoemaker K, Vandebosch A, Sadoff J, Woo W, Cho I, Dunkle LM, Li S, van der Laan L, Gilbert PB, Follmann D, Jaynes H, Kublin JG, Baden LR, Goepfert P, Kotloff K, Gay CL, Falsey AR, El Sahly HM, Sobieszczyk ME, Huang Y, Neuzil KM, Corey L, Grinsztejn B, Gray G, Rouphael N, Luedtke A; COVID-19 Prevention Network CoVPN. Modifiers of COVID-19 vaccine efficacy: Results from four COVID-19 prevention network efficacy trials. Vaccine. 2023 Jul 25;41(33):4899-4906. doi: 10.1016/j.vaccine.2023.06.066. Epub 2023 Jun 23. PMID 37385888
- [Derived] Follmann D, O'Brien MP, Fintzi J, Fay MP, Montefiori D, Mateja A, Herman GA, Hooper AT, Turner KC, Chan KC, Forleo-Neto E, Isa F, Baden LR, El Sahly HM, Janes H, Doria-Rose N, Miller J, Zhou H, Dang W, Benkeser D, Fong Y, Gilbert PB, Marovich M, Cohen MS. Examining protective effects of SARS-CoV-2 neutralizing antibodies after vaccination or monoclonal antibody administration. Nat Commun. 2023 Jun 17;14(1):3605. doi: 10.1038/s41467-023-39292-w. PMID 37330602
- [Derived] Benkeser D, Montefiori DC, McDermott AB, Fong Y, Janes HE, Deng W, Zhou H, Houchens CR, Martins K, Jayashankar L, Castellino F, Flach B, Lin BC, O'Connell S, McDanal C, Eaton A, Sarzotti-Kelsoe M, Lu Y, Yu C, Borate B, van der Laan LWP, Hejazi NS, Kenny A, Carone M, Williamson BD, Garver J, Altonen E, Rudge T, Huynh C, Miller J, El Sahly HM, Baden LR, Frey S, Malkin E, Spector SA, Andrasik MP, Kublin JG, Corey L, Neuzil KM, Carpp LN, Pajon R, Follmann D, Donis RO, Koup RA, Gilbert PB; Immune Assays; Moderna Inc.; Coronavirus Vaccine Prevention Network (CoVPN)/Coronavirus Efficacy (COVE); United States Government (USG)/CoVPN Biostatistics Teams. Comparing antibody assays as correlates of protection against COVID-19 in the COVE mRNA-1273 vaccine efficacy trial. Sci Transl Med. 2023 Apr 19;15(692):eade9078. doi: 10.1126/scitranslmed.ade9078. Epub 2023 Apr 19. PMID 37075127
- [Derived] Chalkias S, Eder F, Essink B, Khetan S, Nestorova B, Feng J, Chen X, Chang Y, Zhou H, Montefiori D, Edwards DK, Girard B, Pajon R, Dutko FJ, Leav B, Walsh SR, Baden LR, Miller JM, Das R. Safety, immunogenicity and antibody persistence of a bivalent Beta-containing booster vaccine against COVID-19: a phase 2/3 trial. Nat Med. 2022 Nov;28(11):2388-2397. doi: 10.1038/s41591-022-02031-7. Epub 2022 Oct 6. PMID 36202997
- [Derived] Fraiman J, Erviti J, Jones M, Greenland S, Whelan P, Kaplan RM, Doshi P. Serious adverse events of special interest following mRNA COVID-19 vaccination in randomized trials in adults. Vaccine. 2022 Sep 22;40(40):5798-5805. doi: 10.1016/j.vaccine.2022.08.036. Epub 2022 Aug 31. PMID 36055877
- [Derived] Follmann D, Janes HE, Buhule OD, Zhou H, Girard B, Marks K, Kotloff K, Desjardins M, Corey L, Neuzil KM, Miller JM, El Sahly HM, Baden LR. Antinucleocapsid Antibodies After SARS-CoV-2 Infection in the Blinded Phase of the Randomized, Placebo-Controlled mRNA-1273 COVID-19 Vaccine Efficacy Clinical Trial. Ann Intern Med. 2022 Sep;175(9):1258-1265. doi: 10.7326/M22-1300. Epub 2022 Jul 5. PMID 35785530
- [Derived] El Sahly HM, Baden LR, Essink B, Montefiori D, McDermont A, Rupp R, Lewis M, Swaminathan S, Griffin C, Fragoso V, Miller VE, Girard B, Paila YD, Deng W, Tomassini JE, Paris R, Schodel F, Das R, August A, Leav B, Miller JM, Zhou H, Pajon R; Coronavirus Efficacy (COVE) Study Group. Humoral Immunogenicity of the mRNA-1273 Vaccine in the Phase 3 Coronavirus Efficacy (COVE) Trial. J Infect Dis. 2022 Nov 11;226(10):1731-1742. doi: 10.1093/infdis/jiac188. PMID 35535503
- [Derived] Pajon R, Paila YD, Girard B, Dixon G, Kacena K, Baden LR, El Sahly HM, Essink B, Mullane KM, Frank I, Denhan D, Kerwin E, Zhao X, Ding B, Deng W, Tomassini JE, Zhou H, Leav B, Schodel F; COVE Trial Consortium. Initial analysis of viral dynamics and circulating viral variants during the mRNA-1273 Phase 3 COVE trial. Nat Med. 2022 Apr;28(4):823-830. doi: 10.1038/s41591-022-01679-5. Epub 2022 Feb 10. PMID 35145311
- [Derived] El Sahly HM, Baden LR, Essink B, Doblecki-Lewis S, Martin JM, Anderson EJ, Campbell TB, Clark J, Jackson LA, Fichtenbaum CJ, Zervos M, Rankin B, Eder F, Feldman G, Kennelly C, Han-Conrad L, Levin M, Neuzil KM, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Polakowski L, Mascola JR, Ledgerwood JE, Graham BS, August A, Clouting H, Deng W, Han S, Leav B, Manzo D, Pajon R, Schodel F, Tomassini JE, Zhou H, Miller J; COVE Study Group. Efficacy of the mRNA-1273 SARS-CoV-2 Vaccine at Completion of Blinded Phase. N Engl J Med. 2021 Nov 4;385(19):1774-1785. doi: 10.1056/NEJMoa2113017. Epub 2021 Sep 22. PMID 34551225
- [Derived] Gilbert PB, Montefiori DC, McDermott A, Fong Y, Benkeser D, Deng W, Zhou H, Houchens CR, Martins K, Jayashankar L, Castellino F, Flach B, Lin BC, O'Connell S, McDanal C, Eaton A, Sarzotti-Kelsoe M, Lu Y, Yu C, Borate B, van der Laan LWP, Hejazi N, Huynh C, Miller J, El Sahly HM, Baden LR, Baron M, De La Cruz L, Gay C, Kalams S, Kelley CF, Kutner M, Andrasik MP, Kublin JG, Corey L, Neuzil KM, Carpp LN, Pajon R, Follmann D, Donis RO, Koup RA. Immune Correlates Analysis of the mRNA-1273 COVID-19 Vaccine Efficacy Trial. medRxiv [Preprint]. 2021 Aug 15:2021.08.09.21261290. doi: 10.1101/2021.08.09.21261290. PMID 34401888
- [Derived] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A participants received mRNA-1273, or placebo. After completion of Part A, participants could have chosen to be unblinded so that participants who received placebo in Part A could request to receive open-label mRNA-1273 in Part B. Eligible participants who received at least one dose of mRNA-1273 in the study had the option to receive a booster dose of mRNA-1273 in Part C.
Groups:
- Part A (Blinded): Placebo: Participants received mRNA-1273-matching placebo on a 2-dose injection schedule (Day 1 and Day 29).
- Part A (Blinded): mRNA-1273: Participants received 100 μg mRNA-1273 on a 2-dose injection schedule (Day 1 and Day 29).
- Part B (Open-label): Placebo: Participants received placebo on a 2-dose injection schedule in Part A and did not receive mRNA-1273 in Part B.
- Part B (Open-label): Placebo/mRNA-1273: Participants received placebo on a 2-dose injection schedule in Part A and received 100 μg mRNA-1273 in Part B.
- Part B (Open-label): mRNA-1273: Participants received mRNA-1273 on a 2-dose injection schedule in Part A and continued follow-up in Part B.
- Part C: mRNA-1273 Booster: Participants received 50 μg mRNA-1273 booster.
Period: Part A: Blinded
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273 | Part B (Open-label): Placebo | Part B (Open-label): Placebo/mRNA-1273 | Part B (Open-label): mRNA-1273 | Part C: mRNA-1273 Booster
Started (Randomization Set (Part A): All participants who were randomized, regardless of the participant's treatment status in the study. Participants were analyzed according to the treatment group to which they were randomized.) | 15206 | 15209 | 0 | 0 | 0 | 0
Received Any Study Injection | 15166 | 15180 | 0 | 0 | 0 | 0
Per-Protocol (PP) Set: (Participants who received any study injection, were severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) negative (defined as no immunologic or virologic evidence of prior COVID-19 at Day 1 before the first dose), and had no major protocol deviations, Participants were analyzed according to the treatment group to which they were randomized. Participants who did not receive the second dose within 21 or 42 days after the first injection date were excluded from the PP Set.) | 14164 | 14287 | 0 | 0 | 0 | 0
Per-Protocol Random Subcohort for Immunogenicity (PPRSI) (All participants in the FAS who were sampled into the random subcohort and received both planned doses (received the treatment the participant was randomized to with Dose 2 received within 21 or 42 days after Dose 1, and no major protocol deviation that impacted critical or key data.) | 272 | 1185 | 0 | 0 | 0 | 0
Solicited Safety Set (All randomized participants who received at least 1 dose and contributed any solicited AR data; (had at least 1 post-baseline solicited safety assessment. Participants were included in the treatment group corresponding to the study vaccination they actually received.) | 15159 | 15179 | 0 | 0 | 0 | 0
Safety Set (All randomized participants who received at least 1 dose. Participants were included in the treatment group corresponding to dose they actually received. For a participant who was randomized to placebo but received any dose of mRNA-1273 at any injection, the participant was included in the mRNA-1273 group in the Safety Set.) | 15162 | 15184 | 0 | 0 | 0 | 0
Full Analysis Set (All randomized participants who received at least 1 dose. Participants were analyzed according to the treatment group to which they were randomized.) | 15166 | 15180 | 0 | 0 | 0 | 0
Completed (Completed Part A (from first dose up to participant decision visit (PDV)/unblinding) and continued to Part B Open-label.) | 14375 | 14661 | 0 | 0 | 0 | 0
Not Completed | 831 | 548 | 0 | 0 | 0 | 0
Not completed — Discontinued from Study in Part A | 831 | 548 | 0 | 0 | 0 | 0
Period: Part B :Open-label
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273 | Part B (Open-label): Placebo | Part B (Open-label): Placebo/mRNA-1273 | Part B (Open-label): mRNA-1273 | Part C: mRNA-1273 Booster
Started (Randomization Set from Part A and who received at least 1 dose. Participants were analyzed according to the treatment group to which they actually received.) | 0 | 0 | 2513 | 12649 | 15184 | 0
Safety Set (All randomized participants who received at least 1 dose in Part A and continued in Part B. Participants were included in the treatment group corresponding to dose they actually received. For a participant who was randomized to placebo but received any dose of mRNA-1273 at any injection, the participant was included in the mRNA-1273 group in the Safety Set.) | 0 | 0 | 2513 | 12649 | 15184 | 0
PP Set (Participants who were randomized in Part A, and were SARS-CoV-2 negative and had no major protocol deviations that impacted critical data.) | 0 | 0 | 2104 | 12060 | 14287 | 0
Participants Who Had PDV/Unblinding) and Had the Option to Receive Booster Dose in Part C | 0 | 0 | 1725 | 12649 | 14661 | 0
Completed (Completed Part B (from first dose up to PDV/unblinding) and had the option to receive booster dose in Part C.) | 0 | 0 | 149 | 10464 | 10171 | 0
Not Completed | 0 | 0 | 2364 | 2185 | 5013 | 0
Not completed — Other than specified | 0 | 0 | 788 | 0 | 523 | 0
Not completed — Discontinued from Study in Part B | 0 | 0 | 1576 | 2185 | 4490 | 0
Period: Part C: Booster
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273 | Part B (Open-label): Placebo | Part B (Open-label): Placebo/mRNA-1273 | Part B (Open-label): mRNA-1273 | Part C: mRNA-1273 Booster
Started (Safety Set: Participants who continued from Part B and opted to receive a booster dose.in Part C.) | 0 | 0 | 0 | 0 | 0 | 19609 (Safety Set: Analysis by treatment received.)
PP Set (Participants who were randomized in Part A, previously receiving 2 doses of mRNA-1273, then received mRNA-1273 booster in Part C, and were pre-booster SARS-CoV-2 negative and had no major protocol deviations that impacted critical data.) | 0 | 0 | 0 | 0 | 0 | 16368
PP Immunogenicity Subset (PPIS) (Participants who were in PPRSI in Part A, randomized and received 2 doses of mRNA-1273 in Part A, were SARS-CoV-2 negative at baseline, received booster in Part C, and had no major protocol deviations that impacted critical data.) | 0 | 0 | 0 | 0 | 0 | 731
PPIS-Negative (Neg) (Participants who were in Part C PPIS and were pre-booster SARS-CoV-2 negative (as determined by non-positive RT-PCR test and negative serology anti-SARS-CoV-2 assay test on or before BD-Day 1).) | 0 | 0 | 0 | 0 | 0 | 682
Completed (Participants are considered to have completed the study if they complete the final visit at Day 759 (Month 25), 24 months following their receipt of the original second dose of investigational product (IP) (where original refers to the IP received following randomization).) | 0 | 0 | 0 | 0 | 0 | 16691
Not Completed | 0 | 0 | 0 | 0 | 0 | 2918
Not completed — Discontinued from Study in Part C | 0 | 0 | 0 | 0 | 0 | 2918

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of treatment.
Groups:
- Placebo: Participants randomized to mRNA-1273-matching placebo and received any study injection in Part A.
- mRNA-1273: Participants randomized to mRNA-1273 and received any study injection in Part A.
- Total: Total of all reporting groups
Arm/Group | Placebo | mRNA-1273 | Total
Number analyzed (Participants) | 15166 | 15180 | 30346
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (15.60) | 51.4 (15.50) | 51.4 (15.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7109 | 7263 | 14372
  Male | 8057 | 7917 | 15974
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3109 | 3121 | 6230
  Not Hispanic or Latino | 11921 | 11917 | 23838
  Unknown or Not Reported | 136 | 142 | 278
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 12001 | 12031 | 24032
  Race: Black or African American | 1531 | 1567 | 3098
  Race: Asian | 739 | 656 | 1395
  Race: American Indian or Alaska Native | 121 | 113 | 234
  Race: Native Hawaiian or other Pacific Islander | 32 | 36 | 68
  Race: Multiracial | 319 | 319 | 638
  Race: Other | 294 | 299 | 593
  Race: Not Reported | 74 | 97 | 171
  Race: Unknown | 55 | 62 | 117

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With a First Occurrence of COVID-19 Starting 14 Days After Second Dose
Description: COVID-19 cases were defined as participants meeting clinical criteria based both on symptoms for COVID-19 and on RT-PCR detection of SARS-CoV-2 from samples collected within 72 hours of the study participant reporting symptoms that met the definition of COVID-19.
  An adjudication committee was assembled for the purpose of reviewing potential cases to determine if the criteria for COVID-19 were met.
Time Frame: From Day 43 (14 days after second dose) up to approximately 7 months after the second dose
Population: Part A PP Set. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 14164 | 14287
Participants | 744 | 55
Statistical Analysis 1: Comparison: Part A (Blinded): Placebo vs Part A (Blinded): mRNA-1273; Vaccine efficacy was defined as the percent reduction in the hazard of the primary endpoint (mRNA-1273 vs. placebo). Null hypothesis of Vaccine Efficacy ≤30%, 95% CI; Test type: Other; p < .0001, Vaccine Efficacy (VE); VE (percent) is demonstrated if the lower limit of the 2-sided confidence interval for the VE is above 30%; VE = 93.2, 95% CI 2-sided [91.0 to 94.8] — VE (percent) was estimated with 1 - Hazard Ratio (mRNA-1273 vs. placebo) from stratified Cox proportional hazard model

2. Primary Outcome: Part A: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) After First Dose
Description: Solicited ARs (local and systemic) were collected in electronic diary (eDiary) within 7 days of dosing. Local ARs included: pain at injection site, erythema (redness) at injection site, swelling/induration (hardness) at injection site, and localized axillary swelling or tenderness ipsilateral to the injection arm. Systemic ARs included: headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, rash, body temperature (potentially fever), and chills. Severity grading for solicited ARs is based on modified Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials. Severity was graded 0-4; a lower score indicated lower severity and a higher score indicated greater severity. The Investigator determined if solicited AR was also to be recorded as an AE. Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is in Reported "Adverse Events" section.
Time Frame: up to Day 7 (7 days after first dose)
Population: Solicited Safety Set: All randomized participants who received at least 1 dose and contributed any solicited AR data; (had at least 1 post-baseline solicited safety assessment. Participants were included in the treatment group corresponding to the study vaccination they actually received. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 15151 | 15166
Participants
  Grade 1 | 5134 | 9329
  Grade 2 | 1782 | 3134
  Grade 3 | 363 | 849
  Grade 4 | 6 | 5

3. Primary Outcome: Part A: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) After Second Dose
Description: Solicited ARs (local and systemic) were collected in eDiary within 7 days of dosing. Local ARs included: pain at injection site, erythema (redness) at injection site, swelling/induration (hardness) at injection site, and localized axillary swelling or tenderness ipsilateral to the injection arm. Systemic ARs included: headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, rash, body temperature (potentially fever), and chills. Severity grading for solicited ARs is based on modified Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials. Severity was graded 0-4; lower score indicated lower severity and a higher score indicated greater severity. The Investigator determined if solicited AR was also to be recorded as an AE. Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is in Reported "Adverse Events" section
Time Frame: Day 29 to Day 35 (from second dose to 7 days after second dose)
Population: Solicited Safety Set: Randomized participants who received at least 1 dose and contributed any solicited AR data. Participants were included in the treatment group corresponding to the study vaccination they actually received. Number analyzed=participants evaluable at specified timepoint. No solicited ARs were collected in Part B because sufficient data had already been captured and analyzed in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 14578 | 14691
Participants
  Grade 1 | 4346 | 4847
  Grade 2 | 1558 | 5800
  Grade 3 | 348 | 2895
  Grade 4 | 3 | 14

4. Primary Outcome: Parts A and B: Number of Participants With Medically Attended AEs (MAAEs) and AEs Leading to Discontinuation
Description: An MAAE is an AE that leads to an unscheduled visit to a healthcare practitioner (HCP). A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Day 1 (after dosing) through end of study (up to Day 759)
Population: Safety Set: All randomized participants who received at least 1 dose. Participants were included in the treatment group corresponding to dose they actually received. For a participant who was randomized to placebo but received any dose of mRNA-1273 at any injection, the participant was included in the mRNA-1273 group in the Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273 | Part B (Open-label): Placebo | Part B (Open-label): Placebo/mRNA-1273 | Part B (Open-label): mRNA-1273
Number analyzed (Participants) | 15162 | 15184 | 2513 | 12649 | 15184
Participants
  MAAEs | 4561 | 3921 | 109 | 5513 | 5809
  AEs Leading to Discontinuation | 25 | 27 | 3 | 30 | 35

5. Primary Outcome: Parts A and B: Number of Participants With Serious AEs (SAEs)
Description: An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Day 1 (after dosing) through end of study (up to Day 759)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273 | Part B (Open-label): Placebo | Part B (Open-label): Placebo/mRNA-1273 | Part B (Open-label): mRNA-1273
Number analyzed (Participants) | 15162 | 15184 | 2513 | 12649 | 15184
Participants | 308 | 292 | 15 | 536 | 516

6. Secondary Outcome: Part A: Number of Participants With Unsolicited AEs up to 28 Days After Any Injection Dose
Description: Unsolicited AE was any AE reported by the participant that was not specified as an AR or was specified as a solicited AR in the protocol but started outside the protocol-defined, post-injection period for reporting solicited ARs. Unsolicited AEs were collected for the 28 days after any injection.
  An AE was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A summary of all SAEs and all nonserious AEs ("Other") reported up to the end of the study, regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to 28 days after any dose
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 15162 | 15184
Participants | 4338 | 4752

7. Secondary Outcome: Parts A and B: Number of Participants With a First Occurrence of Severe COVID-19 Starting 14 Days After Second Dose
Description: COVID-19 cases were defined as participants meeting clinical criteria based on symptoms for COVID-19 and reverse transcriptase polymerase chain reaction (RT-PCR) detection of SARS-CoV-2 from samples collected within 72 hours of the participant reporting symptoms meeting the definition of COVID-19.
  An adjudication committee reviewed potential cases to determine if the criteria for COVID-19 were met.
  Clinical signs indicative of severe COVID-19 systemic illness included any of the following: respiratory rate ≥30 per minute, heart rate ≥125 beats per minute, oxygen saturation (SpO2) ≤93% on room air at sea level, or partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FIO2) <300 millimeter of mercury (mm Hg), or respiratory failure or acute respiratory distress syndrome (ARDS), evidence of shock, or significant acute renal, hepatic, or neurologic dysfunction, or admission to an intensive care unit or death.
Time Frame: From Day 43 (14 days after second dose) up to approximately 8 months for Part A and from PDV/unblinding (at 4 months) to up to 8 months for Part B
Population: Parts A and B PP Sets. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273 | Part B (Open-label): Placebo | Part B (Open-label): Placebo/mRNA-1273 | Part B (Open-label): mRNA-1273
Number analyzed (Participants) | 14164 | 14287 | 2104 | 12060 | 14287
Participants | 106 | 2 | 1 | 8 | 1
Statistical Analysis 1: Comparison: Part A (Blinded): Placebo vs Part A (Blinded): mRNA-1273; Test type: Other; VE; VE = 98.2, 95% CI 2-sided [92.8 to 99.6] — VE (percent) was estimated with 1 - Hazard Ratio (mRNA-1273 vs. placebo) from stratified Cox proportional hazard model

8. Secondary Outcome: Part A: Number of Participants With a First Occurrence of Either COVID-19 or SARS-CoV-2 Infection Regardless of Symptomatology or Severity Starting 14 Days After Second Dose
Description: COVID-19 cases were defined as participants meeting clinical criteria based both on symptoms for COVID-19 and on RT-PCR detection of SARS-CoV-2 from samples collected within 72 hours of the study participant reporting symptoms that met the definition of COVID-19.
  An adjudication committee was assembled for the purpose of reviewing potential cases to determine if the criteria for COVID-19 were met.
  SARS-CoV-2 infection was defined by seroconversion due to infection measured by binding antibody (bAb) levels against SARS-CoV-2 nucleocapsid or by positive RT-PCR at predefined timepoints. Seroconversion was defined by the participant's serostatus at baseline.
Time Frame: From Day 43 (14 days after second dose) up to approximately 7 months after the second dose
Population: Part A PP Set. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 14164 | 14287
Participants | 1339 | 280
Statistical Analysis 1: Comparison: Part A (Blinded): Placebo vs Part A (Blinded): mRNA-1273; Test type: Other; VE = 82.0, 95% CI 2-sided [79.5 to 84.2] — VE (percent) was estimated with 1 - Hazard Ratio (mRNA-1273 vs. placebo) from stratified Cox proportional hazard model

9. Secondary Outcome: Part A: Number of Participants With a Secondary Case Definition of COVID-19 Starting 14 Days After Second Dose
Description: Secondary case definition of COVID-19 was defined as the presence of at least 1 of the following systemic symptoms: fever (temperature
  ≥38ºC), or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle aches or body aches, headache, new loss of taste or smell, sore throat, nasal congestion or rhinorrhea, nausea or vomiting, or diarrhea and a positive nasopharyngeal swab, nasal swab, or saliva sample (or respiratory sample, if hospitalized) for SARS-CoV-2 by RT-PCR.
Time Frame: From Day 43 (14 days after second dose) up to approximately 7 months after the second dose
Population: Part A PP Set. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 14164 | 14287
Participants | 807 | 58
Statistical Analysis 1: Comparison: Part A (Blinded): Placebo vs Part A (Blinded): mRNA-1273; Test type: Other — VE; VE = 93.4, 95% CI 2-sided [91.4 to 94.9] — VE (percent) was estimated with 1 - Hazard Ratio (mRNA-1273 vs. placebo) from stratified Cox proportional hazard model

10. Secondary Outcome: Parts A and B: Number of Participants Who Died Due to a Cause Directly Attributed to a Complication of COVID-19 Starting 14 Days After Second Dose
Time Frame: as for outcome 7
Population: Parts A and B PP Set. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273 | Part B (Open-label): Placebo | Part B (Open-label): Placebo/mRNA-1273 | Part B (Open-label): mRNA-1273
Number analyzed (Participants) | 14164 | 14287 | 2104 | 12060 | 14287
Participants | 3 | 0 | 0 | 0 | 0

11. Secondary Outcome: Part A: Number of Participants With a First Occurrence of COVID-19 Starting 14 Days After First Dose
Description: as for outcome 1
Time Frame: From 14 days after first dose up to approximately 8 months
Population: Part A PP Set. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 14164 | 14287
Participants | 769 | 56
Statistical Analysis 1: Comparison: Part A (Blinded): Placebo vs Part A (Blinded): mRNA-1273; Test type: Other; VE = 93.3, 95% CI 2-sided [91.1 to 94.9] — VE (percent) was estimated with 1 - Hazard Ratio (mRNA-1273 vs. placebo) from stratified Cox proportional hazard model

12. Secondary Outcome: Part A: Number of Participants With a First Occurrence of COVID-19 Starting 14 Days After Second Dose Regardless of Evidence of Prior SARS-CoV-2 Infection
Description: as for outcome 1
Time Frame: From Day 43 (14 days after second dose) up to approximately 7 months after the second dose
Population: Part A FAS. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 15166 | 15180
Participants | 754 | 58
Statistical Analysis 1: Comparison: Part A (Blinded): Placebo vs Part A (Blinded): mRNA-1273; Test type: Other; VE = 82.0, 95% CI 2-sided [79.5 to 84.3] — VE (percent) was estimated with 1 - Hazard Ratio (mRNA-1273 vs. placebo) from stratified Cox proportional hazard model

13. Secondary Outcome: Part A: Number of Participants With a First Occurrence of SARS-CoV-2 Infection in the Absence of Symptoms Defining COVID-19 Starting 14 Days After Second Dose
Description: SARS-CoV-2 infection was defined by seroconversion due to infection measured by binding antibody (bAb) levels against SARS-CoV-2 nucleocapsid or by positive RT-PCR at predefined timepoints. Seroconversion was defined by the participant's serostatus at baseline.
Time Frame: From Day 43 (14 days after second dose) up to approximately 7 months after the second dose
Population: Part A PP Set. Number analyzed=participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 14164 | 14287
Participants | 498 | 214
Statistical Analysis 1: Comparison: Part A (Blinded): Placebo vs Part A (Blinded): mRNA-1273; Test type: Other; VE = 63.0, 95% CI 2-sided [56.6 to 68.5] — VE (percent) was estimated with 1 - Hazard Ratio (mRNA-1273 vs. placebo) from stratified Cox proportional hazard model

14. Secondary Outcome: Part A: Geometric Mean Titer (GMT) of SARS-CoV-2 Specific Neutralizing Antibody (nAb)
Description: GMT (50% inhibitory dose [ID50], 80% inhibitory dose [ID80]) of nAb against SARS-CoV-2 pseudotyped viruses as measured by pseudovirus nAb assay is reported.
  95% CI was based on the t-distribution of log-transformed values for GM titer, then back transformed to original scale for presentation.
  Baseline SARS-CoV-2 Status: Positive if there is immunologic or virologic evidence of prior COVID-19, defined as positive RT-PCR test or positive Elecsys result at Day 1. Negative is defined as negative RT-PCR test and negative Elecsys result at Day 1.
Time Frame: Day 1, Day 29, Day 57
Population: Part A PPRSI Set. Number analyzed=participants evaluable at specified timepoint. Immunogenicity samples from the Part B were not tested and no data were generated as results were not thought to provide additional information.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 272 | 1185
Titer
  Baseline SARS-CoV-2 Negative, ID50, Day 1: number analyzed (Participants) | 142 | 1052
  Baseline SARS-CoV-2 Negative, ID50, Day 1 | NA [NA to NA] — All antibody values were below the lower limit of quantification (LLOQ), therefore, no data for assessment. | 9.624 [9.35 to 9.90]
  Baseline SARS-CoV-2 Negative', ID50, Day 29: number analyzed (Participants) | 142 | 1055
  Baseline SARS-CoV-2 Negative', ID50, Day 29 | 9.515 [9.00 to 10.06] | 54.866 [50.98 to 59.04]
  Baseline SARS-CoV-2 Negative', ID50, Day 57: number analyzed (Participants) | 142 | 1053
  Baseline SARS-CoV-2 Negative', ID50, Day 57 | 9.903 [8.99 to 10.90] | 1081.124 [1019.80 to 1146.14]
  Baseline SARS-CoV-2 Negative', ID80, Day 1: number analyzed (Participants) | 142 | 1052
  Baseline SARS-CoV-2 Negative', ID80, Day 1 | NA [NA to NA] — All antibody values were below LLOQ, therefore, no data for assessment. | 7.332 [7.18 to 7.49]
  Baseline SARS-CoV-2 Negative', ID80, Day 29: number analyzed (Participants) | 142 | 1055
  Baseline SARS-CoV-2 Negative', ID80, Day 29 | 7.279 [7.03 to 7.54] | 19.684 [18.55 to 20.89]
  Baseline SARS-CoV-2 Negative', ID80, Day 57: number analyzed (Participants) | 142 | 1053
  Baseline SARS-CoV-2 Negative', ID80, Day 57 | 7.522 [7.00 to 8.09] | 334.867 [317.84 to 352.81]
  Baseline SARS-CoV-2 Positive, ID50, Day 1: number analyzed (Participants) | 129 | 130
  Baseline SARS-CoV-2 Positive, ID50, Day 1 | 82.519 [59.40 to 114.64] | 68.117 [49.88 to 93.02]
  Baseline SARS-CoV-2 Positive, ID50, Day 29: number analyzed (Participants) | 129 | 130
  Baseline SARS-CoV-2 Positive, ID50, Day 29 | 52.728 [39.45 to 70.48] | 1478.910 [1069.60 to 2044.86]
  Baseline SARS-CoV-2 Positive, ID50, Day 57: number analyzed (Participants) | 130 | 130
  Baseline SARS-CoV-2 Positive, ID50, Day 57 | 47.708 [35.41 to 64.28] | 3145.904 [2539.80 to 3896.66]
  Baseline SARS-CoV-2 Positive, ID80, Day 1: number analyzed (Participants) | 129 | 130
  Baseline SARS-CoV-2 Positive, ID80, Day 1 | 29.580 [22.39 to 39.09] | 24.996 [19.12 to 32.68]
  Baseline SARS-CoV-2 Positive, ID80, Day 29: number analyzed (Participants) | 129 | 130
  Baseline SARS-CoV-2 Positive, ID80, Day 29 | 20.994 [16.42 to 26.84] | 518.388 [380.39 to 706.44]
  Baseline SARS-CoV-2 Positive, ID80, Day 57: number analyzed (Participants) | 130 | 130
  Baseline SARS-CoV-2 Positive, ID80, Day 57 | 19.228 [15.03 to 24.60] | 1099.847 [903.83 to 1338.37]

15. Secondary Outcome: Part A: Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Specific nAb
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants.
  95% CI was calculated based on the difference in the log-transformed values for GMFR, then back transformed to the original scale for presentation. GMFR for ID50 and ID80 neutralizing antibodies against SARS-CoV-2 S-protein, as measured by pseudovirus neutralizing antibody is presented. Baseline SARS-CoV-2 Status: Positive if there is immunologic or virologic evidence of prior COVID-19, defined as positive RT-PCR test or positive Elecsys result at Day 1. Negative is defined as negative RT-PCR test and negative Elecsys result at Day 1
Time Frame: Day 29, Day 57
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 271 | 1182
Ratio
  Baseline SARS-CoV-2 Negative, ID50 Day 29: number analyzed (Participants) | 142 | 1052
  Baseline SARS-CoV-2 Negative, ID50 Day 29 | 1.03 [0.97 to 1.09] | 5.69 [5.29 to 6.12]
  Baseline SARS-CoV-2 Negative, ID50 Day 57: number analyzed (Participants) | 142 | 1050
  Baseline SARS-CoV-2 Negative, ID50 Day 57 | 1.07 [0.97 to 1.18] | 112.30 [105.42 to 119.62]
  Baseline SARS-CoV-2, Negative, ID80 Day 29: number analyzed (Participants) | 142 | 1052
  Baseline SARS-CoV-2, Negative, ID80 Day 29 | 1.02 [0.98 to 1.05] | 2.68 [2.53 to 2.84]
  Baseline SARS-CoV-2 Negative, ID80 Day 57: number analyzed (Participants) | 142 | 1050
  Baseline SARS-CoV-2 Negative, ID80 Day 57 | 1.05 [0.98 to 1.13] | 45.62 [43.21 to 48.17]
  Baseline SARS-CoV-2, Positive, ID50 Day 29: number analyzed (Participants) | 128 | 130
  Baseline SARS-CoV-2, Positive, ID50 Day 29 | 0.64 [0.56 to 0.73] | 21.71 [16.08 to 29.32]
  Baseline SARS-CoV-2 Positive, ID50 Day 57: number analyzed (Participants) | 129 | 130
  Baseline SARS-CoV-2 Positive, ID50 Day 57 | 0.59 [0.50 to 0.69] | 46.18 [34.10 to 62.55]
  Baseline SARS-CoV-2 Positive, ID80 Day 29: number analyzed (Participants) | 128 | 130
  Baseline SARS-CoV-2 Positive, ID80 Day 29 | 0.71 [0.64 to 0.79] | 20.74 [15.30 to 28.10]
  Baseline SARS-CoV-2 Positive, ID80 Day 57: number analyzed (Participants) | 129 | 130
  Baseline SARS-CoV-2 Positive, ID80 Day 57 | 0.66 [0.57 to 0.75] | 44.00 [33.99 to 56.97]

16. Secondary Outcome: Part A: Percentage of Participants With Seroresponse Against SARS-CoV-2
Description: Seroresponse to pseudovirus neutralizing antibody ID50 titer at a participant level is defined as a change from below the LLOQ to equal or above the LLOQ, or at least a 3.3-fold rise if baseline is equal to or above the LLOQ. Seroresponse to pseudovirus neutralizing antibody ID80 titer at a participant level is defined as a change from below the LLOQ to equal or above the LLOQ, or at least a 2.3-fold rise if baseline is equal to or above the LLOQ.
  Baseline SARS-CoV-2 Status: Positive if there is immunologic or virologic evidence of prior COVID-19, defined as positive RT-PCR test or positive Elecsys result at Day 1. Negative is defined as negative RT-PCR test and negative Elecsys result at Day 1.
Time Frame: Day 29, Day 57
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273
Number analyzed (Participants) | 272 | 1185
percentage of participants
  Baseline SARS-CoV-2 Negative, ID50, Day 29: number analyzed (Participants) | 142 | 1055
  Baseline SARS-CoV-2 Negative, ID50, Day 29 | 0.7 [0.0 to 3.9] | 81.4 [78.9 to 83.7]
  Baseline SARS-CoV-2 Negative, ID50, Day 57: number analyzed (Participants) | 142 | 1053
  Baseline SARS-CoV-2 Negative, ID50, Day 57 | 1.4 [0.2 to 5.0] | 98.9 [98.0 to 99.4]
  Baseline SARS-CoV-2 Negative, ID80, Day 29: number analyzed (Participants) | 142 | 1055
  Baseline SARS-CoV-2 Negative, ID80, Day 29 | 0.7 [0.0 to 3.9] | 63.0 [60.0 to 65.9]
  Baseline SARS-CoV-2 Negative, ID80, Day 57: number analyzed (Participants) | 142 | 1053
  Baseline SARS-CoV-2 Negative, ID80, Day 57 | 1.4 [0.2 to 5.0] | 98.9 [98.0 to 99.4]
  Baseline SARS-CoV-2 Positive, ID50, Day 29: number analyzed (Participants) | 129 | 130
  Baseline SARS-CoV-2 Positive, ID50, Day 29 | 0.8 [0.0 to 4.3] | 87.7 [80.8 to 92.8]
  Baseline SARS-CoV-2 Positive, ID50, Day 57: number analyzed (Participants) | 130 | 130
  Baseline SARS-CoV-2 Positive, ID50, Day 57 | 1.6 [0.2 to 5.5] | 94.6 [89.2 to 97.8]
  Baseline SARS-CoV-2 Positive, ID80, Day 29: number analyzed (Participants) | 129 | 130
  Baseline SARS-CoV-2 Positive, ID80, Day 29 | 3.1 [0.9 to 7.8] | 90.0 [83.5 to 94.6]
  Baseline SARS-CoV-2 Positive, ID80, Day 57: number analyzed (Participants) | 130 | 130
  Baseline SARS-CoV-2 Positive, ID80, Day 57 | 2.3 [0.5 to 6.6] | 96.2 [91.3 to 98.7]

17. Secondary Outcome: Part C: GMT of SARS-CoV-2 Specific nAb Measured by Pseudovirus (VAC62)
Description: 95% CI is calculated based on the t-distribution of the log-transformed values for GM value, then back transformed to the original scale for presentation.
Time Frame: Pre-booster (Baseline), post-booster Day 29 and post-booster Day 181
Population: Part C PPIS Set. Number analyzed=participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Part C (Booster): mRNA-1273 Booster: Participants received 50 μg mRNA-1273 booster.
Arm/Group | Part C (Booster): mRNA-1273 Booster
Number analyzed (Participants) | 700
Titer
  Pre-booster (Baseline) | 163.848 [147.977 to 181.421]
  BD Day 29: number analyzed (Participants) | 677
  BD Day 29 | 8122.189 [7603.021 to 8676.808]
  BD Day 181: number analyzed (Participants) | 610
  BD Day 181 | 2951.123 [2701.648 to 3223.636]

18. Secondary Outcome: Part C: Percentage of Participants With Seroresponse Against SARS-CoV-2 Measured by Pseudovirus (VAC62)
Description: Pseudovirus neutralizing antibody (VAC62) from pre-booster is presented. Seroresponse at a participant level is defined as a change from below the LLOQ to >= 4 x LLOQ, or at least a 4-fold rise if pre-booster is equal to or above the LLOQ.
Time Frame: Post-booster Day 29 and post-booster Day 181
Population: Part C PPIS Set. Number analyzed=participants evaluable at specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part C (Booster): mRNA-1273 Booster
Number analyzed (Participants) | 670
percentage of participants
  BD Day 29 | 94.5 [92.5 to 96.1]
  BD Day 181: number analyzed (Participants) | 591
  BD Day 181 | 89.2 [86.4 to 91.6]

19. Secondary Outcome: Part C: Geometric Mean Concentration (GMC) of SARS-CoV-2 Specific nAb After BD Compared to After Second Dose in Part A Measured by Pseudovirus (VAC62)
Description: 95% CI is calculated based on the t-distribution of the log-transformed values for GMC, then back transformed to the original scale for presentation.
Time Frame: Part C BD Day 29 and Part A Day 57
Population: Part C PPIS Set pre-booster SARS-CoV-2 negative. Number analyzed=participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units (AU)/milliliters (mL)
Groups:
- Part A mRNA-1273: Participants received 100 μg mRNA-1273 on a 2-dose injection schedule.
Arm/Group | Part C (Booster): mRNA-1273 Booster | Part A mRNA-1273
Number analyzed (Participants) | 636 | 680
arbitrary units (AU)/milliliters (mL)
  Part C BD Day 29: number analyzed (Participants) | 636 | 0
  Part C BD Day 29 | 7739.680 [7240.926 to 8272.789] |
  Part A Day 57: number analyzed (Participants) | 0 | 680
  Part A Day 57 |  | 1111.274 [1041.684 to 1185.513]
Statistical Analysis 1: Comparison: Part C (Booster): mRNA-1273 Booster vs Part A mRNA-1273; Ratio of GMC 28 days following the booster dose (BD-Day 29) compared with 28 days following second dose (Part A-Day 57); Test type: Non-Inferiority — Non-inferiority of a booster as compared with mRNA-1273 after second dose based on Ratio of GMC is demonstrated if lower bound of 95% CI of Ratio of GMC ≥ 0.67; Ratio of GMC = 6.996, 95% CI 2-sided [6.509 to 7.520]

20. Secondary Outcome: Part C: Percentage of Participants With Seroresponse Against SARS-CoV-2 After BD Compared to After Second Dose in Part A
Description: Pseudovirus neutralizing antibody (VAC62) are presented. Seroresponse at a participant level is defined as a change from below the LLOQ to equal or above 4 x LLOQ, or at least a4-fold rise if baseline (Pre- Dose 1) is equal to or above the LLOQ.
Time Frame: Part C BD Day 29 and Part A Day 57
Population: Part C PPIS Set pre-booster SARS-CoV-2 negative. Number analyzed=participants evaluable at specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part C (Booster): mRNA-1273 Booster | Part A mRNA-1273
Number analyzed (Participants) | 636 | 680
percentage of participants
  Part C BD Day 29: number analyzed (Participants) | 636 | 0
  Part C BD Day 29 | 100 [99.4 to 100] |
  Part A Day 57: number analyzed (Participants) | 0 | 680
  Part A Day 57 |  | 98.8 [97.7 to 99.5]
Statistical Analysis 1: Comparison: Part C (Booster): mRNA-1273 Booster vs Part A mRNA-1273; Seroresponse 28 days following the booster dose (BD-Day 29) compared with 28 days following second dose (Part A-Day 57); Test type: Non-Inferiority — Non-inferiority of a booster as compared with mRNA-1273 after second dose based on SRR difference is demonstrated if lower bound of 95% CI of SRR difference > -10%; Difference in Seroresponse = 0.9, 95% CI 2-sided [0.1 to 1.8] — 95% CI were calculated using adjusted Wald method for the paired binary data

ADVERSE EVENTS:
Time Frame: up to Day 759 (end of study)
Description: All-cause Mortality: Randomized Set for Part A & Safety Sets for Parts B&C.SAEs/"other" AEs: Safety Sets for Parts A&B&C.
  Part A collection: 1st dose to PDV/unblinding/BD/last date observed, whichever was earliest, up to Day 759 Part B collection: PDV/unblinding at 4 months to BD/last date observed, whichever was earliest, up to Day 759 Part C collection: BD through Day 759 Note, not all solicited ARs considered AEs. Investigator determined if solicited AR was also to be recorded as an AE.
Arm/Group | Part A (Blinded): Placebo | Part A (Blinded): mRNA-1273 | Part B (Open-label): Placebo | Part B (Open-label): Placebo/mRNA-1273 | Part B (Open-label): mRNA-1273 | Part C: mRNA-1273 Booster
All-Cause Mortality (participants affected / at risk) | 18/15206 | 16/15209 | 2/2513 | 23/12649 | 35/15184 | 52/19609
Serious Adverse Events (participants affected / at risk) | 308/15162 | 292/15184 | 15/2513 | 536/12649 | 516/15184 | 755/19609
Other Adverse Events (participants affected / at risk) | 2783/15162 | 2247/15184 | 42/2513 | 1739/12649 | 1404/15184 | 8277/19609
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Blinded): Placebo (N=15162) | Part A (Blinded): mRNA-1273 (N=15184) | Part B (Open-label): Placebo (N=2513) | Part B (Open-label): Placebo/mRNA-1273 (N=12649) | Part B (Open-label): mRNA-1273 (N=15184) | Part C: mRNA-1273 Booster (N=19609)
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 3
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Appendiceal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 5 | 4 | 0 | 13 | 7 | 13
Appendicitis perforated (Infections and infestations) | 1 | 1 | 0 | 4 | 4 | 2
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 1
Arthritis gonococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 1
COVID-19 (Infections and infestations) | 33 | 1 | 2 | 10 | 6 | 8
COVID-19 pneumonia (Infections and infestations) | 10 | 0 | 0 | 1 | 4 | 1
Campylobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3 | 0 | 5 | 9 | 8
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Clostridium bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 3 | 0 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Coccidioidomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0
Diverticulitis (Infections and infestations) | 4 | 2 | 0 | 12 | 4 | 6
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fournier's gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Giardiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infected bite (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0
Localised infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Medical device site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 3
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 5 | 2 | 7
Osteomyelitis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 11 | 9 | 1 | 25 | 13 | 19
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 2 | 3 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 6
Postoperative abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 3 | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0 | 0 | 3 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Salpingitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 4 | 4 | 0 | 16 | 9 | 7
Septic encephalopathy (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 4 | 1 | 0 | 3 | 4 | 5
Shigella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Shigella sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Spinal cord infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Streptococcal endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Suspected COVID-19 (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0
Toxic shock syndrome (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 1 | 0 | 8 | 5 | 13
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 4
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2 | 0
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Benign neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 1 | 2
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 2 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 1 | 1
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 1 | 2 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 5 | 5
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 2
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 2 | 2
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 3
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2 | 3 | 1
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1 | 0
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 2
Ovarian clear cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 3 | 4
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 0
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0
Paranasal sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Pleomorphic malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Prolactin-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6 | 0 | 8 | 8 | 7
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 2
Salivary gland cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 1 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
T-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2
Urethral cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2 | 4 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 6 | 3 | 3
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 2 | 3 | 2
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cytokine storm (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 4 | 0 | 0 | 4 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 3 | 0 | 2 | 2 | 6
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 1 | 2 | 4
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 3
Obesity (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3 | 6 | 4
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alcohol use disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 3 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 2 | 3
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 5
Catatonia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 3 | 0 | 3 | 7 | 3
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug dependence (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 2 | 0 | 0 | 1 | 2 | 1
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 1 | 0 | 1 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 2
Schizoaffective disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 2
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Substance use disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Substance-induced mood disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 3 | 0 | 3 | 6 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 0
Alcoholic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Arachnoid cyst (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 1 | 3 | 1
Carotid artery thrombosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 6 | 0 | 7 | 8 | 12
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 4
Drug withdrawal convulsions (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 2 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemiplegic migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 4
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Idiopathic partial epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Incoherent (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Lacunar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 2 | 1 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2
Multiple sclerosis (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 3
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 4
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 1 | 3 | 0 | 0 | 3 | 6
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Stiff person syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 3 | 0 | 1 | 2 | 1
Syncope (Nervous system disorders) | 7 | 6 | 0 | 4 | 10 | 13
Thalamic infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2
Transient global amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 0 | 4 | 2 | 13
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vestibular migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 1 | 1 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac disorders (Ear and labyrinth disorders) | 45 | 44 | 2 | 85 | 81 | 142
Acute coronary syndrome (Ear and labyrinth disorders) | 0 | 3 | 0 | 3 | 0 | 5
Acute left ventricular failure (Ear and labyrinth disorders) | 2 | 1 | 0 | 4 | 2 | 0
Acute myocardial infarction (Ear and labyrinth disorders) | 6 | 4 | 1 | 10 | 11 | 21
Angina pectoris (Ear and labyrinth disorders) | 1 | 3 | 0 | 3 | 8 | 5
Angina unstable (Ear and labyrinth disorders) | 0 | 1 | 0 | 6 | 1 | 3
Aortic valve incompetence (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 2 | 0
Aortic valve stenosis (Ear and labyrinth disorders) | 0 | 0 | 0 | 4 | 0 | 1
Arrhythmia (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 1
Arteriosclerosis coronary artery (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arteriospasm coronary (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Ear and labyrinth disorders) | 11 | 7 | 0 | 11 | 13 | 27
Atrial flutter (Ear and labyrinth disorders) | 2 | 2 | 0 | 5 | 4 | 5
Atrial tachycardia (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0
Atrioventricular block (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block complete (Ear and labyrinth disorders) | 1 | 0 | 0 | 2 | 0 | 4
Atrioventricular block second degree (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 3 | 2
Bundle branch block left (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bundle branch block right (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 5 | 9
Cardiac disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Ear and labyrinth disorders) | 2 | 1 | 1 | 3 | 1 | 1
Cardiac failure acute (Ear and labyrinth disorders) | 1 | 1 | 0 | 3 | 1 | 3
Cardiac failure chronic (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Ear and labyrinth disorders) | 4 | 4 | 1 | 8 | 10 | 10
Cardiac flutter (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Ear and labyrinth disorders) | 1 | 2 | 0 | 0 | 0 | 1
Cardiogenic shock (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 4
Cardiomegaly (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiomyopathy (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2 | 0
Cardiopulmonary failure (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiovascular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2
Chronic left ventricular failure (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Ear and labyrinth disorders) | 3 | 5 | 0 | 15 | 12 | 18
Coronary artery insufficiency (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery occlusion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 3 | 0
Coronary artery stenosis (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular failure (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 0 | 1
Microvascular coronary artery disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1 | 0
Mitral valve prolapse (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mitral valve stenosis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Ear and labyrinth disorders) | 10 | 8 | 0 | 6 | 8 | 14
Myocardial ischaemia (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2
Palpitations (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Paroxysmal atrioventricular block (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 1
Pericarditis (Ear and labyrinth disorders) | 3 | 2 | 0 | 0 | 0 | 2
Pulseless electrical activity (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0
Sinoatrial block (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus node dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 2
Sinus tachycardia (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0 | 1
Stress cardiomyopathy (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 2 | 0
Supraventricular tachycardia (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 1 | 2
Tachycardia (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ventricular arrhythmia (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 1 | 0
Ventricular fibrillation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Ear and labyrinth disorders) | 0 | 0 | 0 | 4 | 0 | 2
Aortic aneurysm (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aortic disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 3 | 0 | 0 | 2 | 2 | 2
Arterial haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 4 | 0 | 2 | 7 | 7
Embolism venous (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fibromuscular dysplasia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 2 | 2 | 0 | 5 | 1 | 3
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 3
Hypertensive emergency (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypertensive urgency (Vascular disorders) | 1 | 2 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0 | 2 | 4 | 8
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
May-Thurner syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 4
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 3 | 1 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Polyarteritis nodosa (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 0 | 5 | 6 | 6
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 2 | 3
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 1 | 5 | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 3 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 3 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 5 | 2 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 3 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 0 | 11 | 11 | 16
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 1 | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cannabinoid hyperemesis syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 4 | 4 | 0 | 1 | 0 | 4
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 2
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastric fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 4 | 0 | 4 | 3 | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1 | 4
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 0 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Internal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 4 | 6
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 1 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 4 | 4 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 1 | 4
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 3 | 0 | 4 | 4 | 10
Terminal ileitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tooth socket haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 3 | 0 | 5 | 6 | 8
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 4 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 2 | 4 | 1
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis of pregnancy (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders (Hepatobiliary disorders) | 2 | 2 | 0 | 2 | 0 | 5
Acute generalised exanthematous pustulosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 1
Decubitus ulcer (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis bullous (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug eruption (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythema nodosum (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Excessive skin (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash vesicular (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 3 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 4 | 0 | 5
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 3 | 2 | 2
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4 | 3 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 2 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 | 12 | 1 | 30 | 21 | 21
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2 | 2 | 4
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 2 | 1 | 2
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 3 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 6 | 0 | 7 | 10 | 9
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 3 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 5 | 0 | 11 | 3 | 7
Renal aneurysm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 1 | 3
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 3 | 2 | 4
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 2 | 0 | 6 | 5 | 8
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 3 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0 | 2 | 5 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 1 | 0
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 3
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Congenital, familial and genetic disorders (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 2 | 0
Arnold-Chiari malformation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0
Talipes (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitello-intestinal duct remnant (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 6 | 1 | 3
Death (General disorders) | 2 | 2 | 0 | 2 | 3 | 7
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Incarcerated hernia (General disorders) | 2 | 0 | 0 | 0 | 1 | 1
Medical device pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 5 | 0 | 3 | 6 | 5
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Procedural failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 3
Strangulated hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Swelling face (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 3 | 0 | 0 | 0 | 2 | 0
Vascular stent stenosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Investigations (General disorders) | 1 | 4 | 0 | 4 | 4 | 6
Ammonia increased (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anticoagulation drug level above therapeutic (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Ejection fraction decreased (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Heart rate decreased (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Heart rate irregular (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hepatic enzyme increased (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hormone level abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Liver function test increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial necrosis marker increased (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Platelet count decreased (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Weight increased (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 2
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 3 | 2 | 6
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Central cord syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 3 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 2 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 2 | 0 | 3 | 1 | 9
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 4
Femur fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 5 | 2 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 3
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 2 | 1 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Immunisation anxiety related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Open globe injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 3 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2
Pelvic bone injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 2
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 3
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1 | 2 | 5
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 3 | 1 | 7
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 3
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 2 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 2
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 3 | 1 | 3
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 3 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 2
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 3
Ureteric injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 3
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 2
Abdominoplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Liposuction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Mammoplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Social circumstances (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1 | 0
Physical assault (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Sexual abuse (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Product issues (Surgical and medical procedures) | 1 | 0 | 0 | 3 | 0 | 1
Device dislocation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Device electrical impedance issue (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Device failure (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Device loosening (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Lead dislodgement (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Blinded): Placebo (N=15162) | Part A (Blinded): mRNA-1273 (N=15184) | Part B (Open-label): Placebo (N=2513) | Part B (Open-label): Placebo/mRNA-1273 (N=12649) | Part B (Open-label): mRNA-1273 (N=15184) | Part C: mRNA-1273 Booster (N=19609)
COVID-19 (Infections and infestations) | 947 | 92 | 21 | 489 | 650 | 4885
Upper respiratory tract infection (Infections and infestations) | 361 | 305 | 18 | 441 | 491 | 1017
Headache (Nervous system disorders) | 1046 | 1087 | 4 | 384 | 200 | 1150
Fatigue (General disorders) | 954 | 1078 | 6 | 343 | 141 | 1515
Injection site pain (General disorders) | 165 | 327 | 0 | 559 | 45 | 2764

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT04470427/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT04470427/SAP_001.pdf
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT04470427/ICF_002.pdf